CLINICAL TRIAL: NCT01673178
Title: A Phase 1, Placebo-controlled, Randomized Trial To Assess The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of Multiple Iv Doses Of Pf-05231023 In Obese Hyperlipidemic Adult Subjects With And Without Type 2 Diabetes Mellitus On A Background Of Atorvastatin
Brief Title: Multiple Dose Study Of PF-05231023 In Adult Subjects Who Have Poor Lipid Control With And Without Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B2901011
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Results first posted 2015-01-14 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes Melliuts, Type 2
Keywords: Type 2 diabetes; safety; multiple dose; intravenous
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — PF-05231023

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo Arm (Placebo Comparator)
  Interventions: Other: Placebo
- 25 mg (Experimental)
  Interventions: Drug: 25 mg PF-05231023
- 50 mg (Experimental)
  Interventions: Drug: 50 mg PF-05231023
- 100 mg (Experimental)
  Interventions: Drug: 100 mg PF-05231023
- 150 mg (Experimental)
  Interventions: Drug: 150 mg PF-05231023

INTERVENTIONS:
Other: Placebo — 0.9% w/v sodium chloride injection, United States Pharmacopeia (USP), once a week for 4 weeks
  Arms: Placebo Arm
Drug: 25 mg PF-05231023 — 25 mg IV once a week for 4 weeks
  Arms: 25 mg
Drug: 50 mg PF-05231023 — 50 mg IV once a week for 4 weeks
  Arms: 50 mg
Drug: 100 mg PF-05231023 — 100 mg IV once a week for 4 weeks
  Arms: 100 mg
Drug: 150 mg PF-05231023 — 150 mg IV once a week for 4 weeks
  Arms: 150 mg

SUMMARY:
This is a trial in obese subjects who have poor lipid control with and without Type 2 diabetes mellitus to study the safety, tolerability and pharmacokinetics of multiple doses of PF-05231023

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects of non-childbearing potential between the ages of 30 and 70 years with and without a diagnosis of Type 2 diabetes mellitus (according to the American Diabetes Association guidelines).
* Subjects with poor lipid control as confirmed by laboratory tests.
* BMI of 30 to 40 Kg/m2 and a total body weight of >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding asymptomatic, seasonal allergies at time of dosing).
* Levels of blood enzymes indicating pancreatitis or elevated liver function enzymes outside of the laboratory's reference range as confirmed by laboratory tests.
* Subjects with Type 1 Diabetes Mellitus.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2012-10; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (17):
- United States (17):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Profil Institute for Clinical Research, Inc., Chula Vista, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Avail Clinical Research, LLC, DeLand, Florida
  - Elite Research Institute, Miami, Florida
  - Miami Research Associates, Inc., South Miami, Florida
  - MRA Clinical Research, LLC, South Miami, Florida
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - L-MARC Research Center, Louisville, Kentucky
  - Prism Research, Saint Paul, Minnesota
  - High Point Clinical Trials Center, LLC, High Point, North Carolina
  - Carolina Phase 1 Research, Raleigh, North Carolina
  - Wake Internal Medicine Consultants, Raleigh, North Carolina
  - Medpace Clinical Pharmacology Unit, Cincinnati, Ohio
  - Community Research, Cincinnati, Ohio
  - Mercy Hospital Pharmacy, Cincinnati, Ohio
  - Covance Clinical Research Unit, Dallas, Texas

REFERENCES:
- [Derived] Kim AM, Somayaji VR, Dong JQ, Rolph TP, Weng Y, Chabot JR, Gropp KE, Talukdar S, Calle RA. Once-weekly administration of a long-acting fibroblast growth factor 21 analogue modulates lipids, bone turnover markers, blood pressure and body weight differently in obese people with hypertriglyceridaemia and in non-human primates. Diabetes Obes Metab. 2017 Dec;19(12):1762-1772. doi: 10.1111/dom.13023. Epub 2017 Jul 21. PMID 28573777
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2901011&StudyName=Multiple%20Dose%20Study%20Of%20PF-05231023%20In%20Adult%20Subjects%20Who%20Have%20Poor%20Lipid%20Control%20With%20And%20Without%20Type%202%20Diabetes%20Mellitus

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo matched to PF-05231023 intravenous infusion over 30 minutes once weekly up to Week 4.
- PF-05231023 25 mg: PF-05231023 25 milligram (mg) intravenous infusion over 30 minutes once weekly up to Week 4.
- PF-05231023 50 mg: PF-05231023 50 mg intravenous infusion over 30 minutes once weekly up to Week 4.
- PF-05231023 100 mg: PF-05231023 100 mg intravenous infusion over 30 minutes once weekly up to Week 4.
- PF-05231023 150 mg: PF-05231023 150 mg intravenous infusion over 30 minutes once weekly up to Week 4.
Period: Overall Study
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Started | 22 | 21 | 21 | 22 | 21
Completed | 19 | 19 | 18 | 14 | 19
Not Completed | 3 | 2 | 3 | 8 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 4 | 2
Not completed — Protocol Violation | 1 | 1 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 2 | 0
Not completed — Other | 1 | 0 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis set included all participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg | Total
Number analyzed (Participants) | 22 | 21 | 21 | 22 | 21 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (8.0) | 54.6 (8.3) | 53.4 (9.5) | 53.0 (7.4) | 53.2 (8.0) | 53.4 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 4 | 5 | 4 | 31
  Male | 11 | 14 | 17 | 17 | 17 | 76

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent events were between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Baseline up to 28 days after last dose
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 22 | 21 | 21 | 22 | 21
participants
  AEs | 11 | 15 | 10 | 13 | 12
  SAEs | 1 | 2 | 0 | 1 | 0

2. Primary Outcome: Number of Participants With Laboratory Abnormalities
Description: Criteria for laboratory test abnormality: Hematology (hemoglobin, hematocrit, red blood corpuscles [RBC] count: less than [<]0.8*lower limit of normal [LLN], platelets: <0.5*LLN/greater than [>]1.75*upper limit of normal [ULN], leukocytes: <0.6*LLN or >1.5*ULN, lymphocytes, total neutrophils: <0.8*LLN or >1.2*ULN, basophils, eosinophil: <0.8*LLN, monocytes: >1.2*ULN); Liver Function (aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase: >0.3*ULN, total protein, albumin: <0.8*LLN or >1.2*ULN); total bilirubin, direct bilirubin, indirect bilirubin: >1.5*ULN; Renal Function (blood urea nitrogen, creatinine: >1.3*ULN, uric acid: >1.2*ULN); Electrolytes (sodium: <0.95*LLN or >1.05*ULN, potassium, chloride, calcium, bicarbonate: <0.9*LLN or >1.1*ULN; creatine kinase: >2.0*ULN; glucose fasting: <0.6*LLN or >1.5*ULN, urine white blood corpuscles [WBC] and RBC: greater than or equal to (>=) 20/High Power Field [HPF]).
Time Frame: Baseline up to Day 49
Population: Safety analysis set included all participants who received at least 1 dose of study medication. Here "N" (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 22 | 21 | 21 | 20 | 21
participants | 18 | 17 | 17 | 12 | 15

3. Primary Outcome: Number of Participants With Clinically Significant Vital Sign Abnormalities
Description: Criteria for clinically significant vital signs abnormalities included supine/sitting pulse rate of <40 beats per minute (bpm) or >120 bpm, supine systolic blood pressure (SBP) of <90 millimeter of mercury (mmHg), >=30 mmHg maximum increase and decrease from baseline in same posture, supine diastolic blood pressure (DBP) of <50 mmHg; >=20 mmHg maximum increase and decrease from baseline in same posture.
Time Frame: Baseline up to Day 49
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 22 | 21 | 21 | 22 | 21
participants
  Supine SBP: <90 mmHg | 1 | 1 | 0 | 0 | 0
  Supine DBP: <50 mmHg | 0 | 0 | 1 | 0 | 0
  Maximum Increase in Supine SBP: >=30 mmHg | 1 | 5 | 4 | 6 | 2
  Maximum Increase in Supine DBP: >=20 mmHg | 2 | 4 | 3 | 1 | 2
  Maximum Decrease in Supine SBP: >=30 mmHg | 3 | 2 | 2 | 0 | 0
  Maximum Decrease in Supine DBP: >=20 mmHg | 5 | 1 | 4 | 4 | 2
  Supine Pulse Rate: <40 bpm | 0 | 0 | 0 | 0 | 0
  Supine Pulse Rate: >120 bpm | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Electrocardiogram Findings
Description: Clinically significant ECG findings included PR interval >=300 milliseconds (msec) or >=25 percent (%) increase from baseline (if baseline PR interval >200 msec) or >=50% increase (if baseline PR interval less than or equal to [<=] 200 msec); QRS interval >=140 msec or >=50% increase from baseline; QT interval >=500 msec, corrected QT interval based on Fridericia's formula (QTcF) 450 to <480 msec, 480 to <500 msec, >=500 msec or >=30 msec but <60 msec increase from baseline or >=60 msec increase from baseline.
Time Frame: Baseline up to Day 49
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 22 | 21 | 21 | 22 | 21
participants
  Maximum PR interval: >=300 msec | 0 | 0 | 0 | 0 | 0
  Maximum PR interval increase : 25% or 50% | 0 | 0 | 0 | 0 | 0
  Maximum QRS complex: >=140 msec | 0 | 0 | 0 | 0 | 0
  Maximum QRS complex increase from baseline:>=50% | 0 | 0 | 0 | 0 | 0
  Maximum QT interval: >=500 msec | 0 | 0 | 0 | 0 | 0
  Maximum QTcF interval: 450-<480 msec | 4 | 3 | 3 | 1 | 3
  Maximum QTcF interval: 480-<500 msec | 0 | 0 | 0 | 0 | 0
  Maximum QTcF interval: >=500 msec | 0 | 0 | 0 | 0 | 0
  Maximum QTcF interval increase: >= 30 to <60 msec | 7 | 4 | 1 | 1 | 4
  Maximum QTCF interval increase: >=60 msec | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Abnormal Physical Examinations
Description: Physical examination included general examination and examination of head, ears, eyes, nose, mouth, throat, neck, abdomen, skin, heart, lungs, lymph nodes, and gastrointestinal and musculoskeletal and neurological system.
Time Frame: Baseline up to Day 49
Population: Physical examination data reported in this study was for identification of adverse events and were reported as an adverse event in the adverse event section.
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Thyroid Stimulating Hormone (TSH) Level at Baseline
Description: Results are reported in micro international units per milliliter (mcIU/mL).
Time Frame: Baseline
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: mcIU/mL
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 22 | 21 | 21 | 22 | 21
mcIU/mL | 1.57 (0.65) | 2.14 (1.25) | 1.96 (1.06) | 1.88 (1.02) | 2.06 (0.87)

7. Primary Outcome: Thyroid Stimulating Hormone (TSH) Level at Day 1
Time Frame: Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcIU/mL
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 22 | 21 | 21 | 21 | 21
mcIU/mL | 1.96 (0.95) | 2.19 (1.10) | 2.40 (1.40) | 2.26 (1.27) | 4.21 (6.67)

8. Primary Outcome: Thyroid Stimulating Hormone (TSH) Level at Day 25
Time Frame: Day 25
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcIU/mL
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 19 | 20 | 18 | 15 | 19
mcIU/mL | 2.70 (3.68) | 2.13 (1.07) | 2.43 (0.87) | 2.52 (1.38) | 4.06 (5.69)

9. Primary Outcome: Thyroid Stimulating Hormone (TSH) Level at Day 39
Time Frame: Day 39
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcIU/mL
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 18 | 19 | 18 | 14 | 19
mcIU/mL | 3.69 (8.11) | 2.08 (1.54) | 2.17 (1.12) | 2.50 (1.37) | 3.10 (3.28)

10. Primary Outcome: Thyroid Stimulating Hormone (TSH) Level at Day 49
Time Frame: Day 49
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcIU/mL
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 18 | 19 | 18 | 14 | 18
mcIU/mL | 3.42 (7.45) | 1.98 (1.16) | 2.43 (1.78) | 2.55 (1.06) | 3.10 (2.03)

11. Primary Outcome: Phosphate Level at Baseline
Time Frame: Baseline
Population: as for outcome 2
Measure: Median (Full Range); unit: milligram per deciliter (mg/dL)
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 22 | 21 | 20 | 22 | 21
milligram per deciliter (mg/dL) | 4.1 [3.0 to 5.1] | 3.8 [3.1 to 5.0] | 3.9 [3.0 to 5.3] | 4.0 [3.0 to 5.2] | 4.0 [2.9 to 4.5]

12. Primary Outcome: Change From Baseline in Phosphate Level at Day 8
Time Frame: Baseline, Day 8
Population: as for outcome 2
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 22 | 20 | 20 | 17 | 19
mg/dL | -0.2 [-1.4 to 0.8] | -0.4 [-1.4 to 0.6] | 0.1 [-0.8 to 0.6] | 0.0 [-1.0 to 0.8] | -0.3 [-1.0 to 1.0]

13. Primary Outcome: Change From Baseline in Phosphate Level at Day 15
Time Frame: Baseline, Day 15
Population: as for outcome 2
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 19 | 20 | 16 | 17 | 20
mg/dL | -0.2 [-1.2 to 0.8] | -0.2 [-2.3 to 0.7] | 0.2 [-1.6 to 1.3] | -0.1 [-0.9 to 0.9] | -0.2 [-0.8 to 0.5]

14. Primary Outcome: Change From Baseline in Phosphate Level at Day 25
Time Frame: Baseline, Day 25
Population: as for outcome 2
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 19 | 20 | 17 | 15 | 19
mg/dL | -0.1 [-1.1 to 0.8] | -0.2 [-1.1 to 0.5] | 0.2 [-0.6 to 1.1] | 0.1 [-0.6 to 0.8] | 0.0 [-0.7 to 0.4]

15. Primary Outcome: Change From Baseline in Phosphate Level at Day 49
Time Frame: Baseline, Day 49
Population: as for outcome 2
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 19 | 19 | 17 | 14 | 19
mg/dL | -0.40 [-1.50 to 0.30] | -0.40 [-1.40 to 1.00] | -0.20 [-1.20 to 1.20] | -0.30 [-1.10 to 0.70] | -0.10 [-0.90 to 0.90]

16. Primary Outcome: Creatine Phosphokinase (CPK) Level at Baseline
Time Frame: Baseline
Population: as for outcome 2
Measure: Median (Full Range); unit: units per liter (U/L)
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 22 | 21 | 20 | 22 | 21
units per liter (U/L) | 73 [26 to 471] | 94 [42 to 493] | 94 [38 to 399] | 103 [45 to 699] | 108 [44 to 173]

17. Primary Outcome: Change From Baseline in Creatine Phosphokinase (CPK) Level at Day 8
Time Frame: Baseline, Day 8
Population: as for outcome 2
Measure: Median (Full Range); unit: U/L
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 22 | 20 | 20 | 17 | 19
U/L | 10 [-260 to 143] | 32 [-21 to 850] | 13 [-70 to 245] | 25 [-175 to 92] | 13 [-27 to 7614]

18. Primary Outcome: Change From Baseline in Creatine Phosphokinase (CPK) Level at Day 15
Time Frame: Baseline, Day 15
Population: as for outcome 2
Measure: Median (Full Range); unit: U/L
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 19 | 20 | 16 | 16 | 20
U/L | 28 [-34 to 852] | 20 [-34 to 629] | 7 [-97 to 243] | 22 [-113 to 238] | 18 [-62 to 248]

19. Primary Outcome: Change From Baseline in Creatine Phosphokinase (CPK) Level at Day 25
Time Frame: Baseline, Day 25
Population: as for outcome 2
Measure: Median (Full Range); unit: U/L
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 18 | 19 | 16 | 15 | 18
U/L | -5 [-246 to 32] | -6 [-38 to 48] | -15 [-110 to 19] | -8 [-54 to 771] | -3 [-90 to 39]

20. Primary Outcome: Change From Baseline in Creatine Phosphokinase (CPK) Level at Day 49
Time Frame: Baseline, Day 49
Population: as for outcome 2
Measure: Median (Full Range); unit: U/L
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 19 | 19 | 17 | 14 | 19
U/L | 21 [-141 to 2214] | 40 [-30 to 494] | 27 [-85 to 292] | 43 [-16 to 216] | 10 [-62 to 139]

21. Primary Outcome: Serum N-terminal Propeptides of Type 1 Collagen (PINP) and C-Telopeptide Cross-Linking of Type 1 Collagen (CTX) Levels at Baseline
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (NG/ML)
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 22 | 21 | 21 | 21 | 21
nanogram per milliliter (NG/ML)
  PINP | 46.3 (15.6) | 41.7 (17.0) | 44.7 (19.4) | 45.0 (19.8) | 44.6 (17.6)
  CTX | 0.35 (0.11) | 0.33 (0.16) | 0.35 (0.15) | 0.38 (0.20) | 0.37 (0.19)

22. Primary Outcome: Percent Change From Baseline in Serum N-terminal Propeptides of Type 1 Collagen (PINP) and C-Telopeptide Cross-Linking of Type 1 Collagen (CTX) Levels at Day 25
Time Frame: Baseline, Day 25
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 19 | 20 | 18 | 15 | 19
percent change
  PINP | -0.8 (13.5) | -14.5 (11.0) | -13.4 (13.3) | -17.6 (12.8) | -19.8 (9.2)
  CTX | 5.2 (15.5) | 2.3 (19.7) | 8.0 (23.6) | 7.3 (17.7) | 7.9 (19.4)

23. Primary Outcome: Percent Change From Baseline in Serum N-terminal Propeptides of Type 1 Collagen (PINP) and C-Telopeptide Cross-Linking of Type 1 Collagen (CTX) Levels at Day 39
Time Frame: Baseline, Day 39
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 18 | 19 | 18 | 14 | 19
percent change
  PINP | -2.8 (13.6) | -9.8 (12.4) | -6.6 (15.6) | -10.3 (12.8) | -11.0 (13.5)
  CTX | -7.3 (21.7) | -4.2 (21.1) | -3.5 (20.2) | -13.1 (18.2) | -3.0 (31.5)

24. Primary Outcome: Percent Change From Baseline Serum N-terminal Propeptides of Type 1 Collagen (PINP) and C-Telopeptide Cross-Linking of Type 1 Collagen (CTX) Levels at Day 49
Time Frame: Baseline, Day 49
Population: Safety analysis set included all participants who receive at least 1 dose of study medication. Here "N" (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 18 | 19 | 18 | 14 | 18
percent change
  PINP | -3.0 (16.4) | -9.4 (16.9) | -1.3 (20.3) | -4.6 (15.0) | -7.4 (18.3)
  CTX | 1.5 (20.8) | 7.5 (30.9) | -3.9 (33.8) | -16.6 (15.3) | -5.3 (25.0)

25. Primary Outcome: Blood Osteocalcin and Bone-Specific Alkaline Phosphatase Levels at Baseline
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: microgram per liter (mcg/l)
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 22 | 21 | 21 | 21 | 21
microgram per liter (mcg/l)
  Blood Osteocalcin | 18.8 (5.4) | 19.2 (5.9) | 18.5 (6.3) | 20.2 (8.2) | 19.9 (7.0)
  Bone-Specific Alkaline Phosphatase | 13.0 (5.7) | 11.7 (3.9) | 11.2 (4.8) | 10.0 (3.0) | 11.2 (4.2)

26. Primary Outcome: Percent Change From Baseline in Blood Osteocalcin and Bone-Specific Alkaline Phosphatase Levels at Day 25
Time Frame: Baseline, Day 25
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 19 | 20 | 18 | 15 | 19
percent change
  Blood Osteocalcin | -2.4 (8.2) | -12.2 (9.6) | -6.4 (14.0) | -7.1 (11.2) | -4.8 (8.2)
  Bone-Specific Alkaline Phosphatase | -4.3 (14.5) | -6.6 (17.0) | -0.4 (15.4) | -5.1 (16.2) | -7.1 (13.1)

27. Primary Outcome: Percent Change From Baseline in Blood Osteocalcin and Bone-Specific Alkaline Phosphatase Levels at Day 39
Time Frame: Baseline, Day 39
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 18 | 19 | 18 | 14 | 19
percent change
  Blood Osteocalcin | -1.8 (12.6) | -10.7 (9.1) | -11.6 (12.4) | -14.7 (11.6) | -13.4 (13.3)
  Bone-Specific Alkaline Phosphatase | -5.0 (20.7) | -5.1 (11.2) | 3.0 (18.9) | -13.0 (19.0) | -8.1 (12.4)

28. Primary Outcome: Percent Change From Baseline in Blood Osteocalcin and Bone-Specific Alkaline Phosphatase Levels at Day 49
Time Frame: Baseline, Day 49
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 18 | 19 | 18 | 14 | 18
percent change
  Blood Osteocalcin | -4.5 (11.9) | -10.7 (8.5) | -5.1 (17.1) | -11.0 (9.3) | -4.8 (12.3)
  Bone-Specific Alkaline Phosphatase | -3.8 (20.6) | -3.9 (14.4) | -0.9 (13.2) | -9.6 (16.6) | 0.7 (27.1)

29. Primary Outcome: Tartrate-resistant Acid Phosphatase Isoform 5b (TRAP 5b) Levels at Baseline
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 21 | 21 | 21 | 21 | 21
units per liter (U/L) | 2.97 (0.53) | 2.72 (0.48) | 3.10 (0.73) | 2.78 (0.62) | 3.08 (0.65)

30. Primary Outcome: Percent Change From Baseline in Tartrate-resistant Acid Phosphatase Isoform 5b (TRAP 5b) Levels at Day 25
Time Frame: Baseline, Day 25
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 18 | 20 | 18 | 15 | 19
percent change | 1.3 (9.4) | -1.7 (12.6) | 1.9 (11.0) | -0.4 (10.6) | -1.4 (10.9)

31. Primary Outcome: Percent Change From Baseline in Tartrate-resistant Acid Phosphatase Isoform 5b (TRAP 5b) Levels at Day 39
Time Frame: Baseline, Day 39
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 17 | 19 | 18 | 14 | 19
percent change | 0.5 (10.7) | -0.4 (11.6) | 0.2 (10.0) | -2.9 (9.9) | 3.7 (16.2)

32. Primary Outcome: Percent Change From Baseline in Tartrate-resistant Acid Phosphatase Isoform 5b (TRAP 5b) Levels at Day 49
Time Frame: Day 49
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 17 | 19 | 18 | 14 | 18
percent change | -2.4 (10.2) | 3.1 (18.0) | -0.8 (12.0) | -0.1 (9.3) | -1.1 (15.8)

33. Primary Outcome: Average Urinary Calcium and Phosphate Levels Over 24 Hours at Baseline
Time Frame: Baseline
Population: Safety analysis set included all participants who received at least 1 dose of study medication. Here "n" signifies those participants who were evaluable for this measure at specified time-points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: milligram per 24 hours (mg/24hr)
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 22 | 21 | 21 | 22 | 21
milligram per 24 hours (mg/24hr)
  Urine Calcium (n=20, 20, 20, 20, 21) | 296.4 (143.4) | 202.1 (104.5) | 224.3 (122.2) | 205.3 (100.1) | 207.4 (112.9)
  Urine Phosphate (n=21, 20, 20, 21, 21) | 922.1 (430.3) | 673.2 (228.3) | 859.1 (318.7) | 795.4 (294.4) | 755.3 (292.1)

34. Primary Outcome: Change From Baseline in Average Urinary Calcium and Phosphate Levels Over 24 Hours at Day 24
Time Frame: Day 24
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: mg/24 hours
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 22 | 21 | 21 | 22 | 21
mg/24 hours
  Urine Calcium (n=17, 17, 16, 15, 19) | -29.3 (106.3) | -9.1 (69.6) | 38.0 (131.9) | 8.2 (69.0) | 5.1 (89.7)
  Urine Phosphate (n=18, 16, 16, 15, 18) | 18.8 (276.0) | 225.8 (283.4) | 241.6 (436.0) | 244.1 (363.4) | 484.4 (514.7)

35. Primary Outcome: Number of Participants With Anti-PF-05231023 Antibodies and Neutralizing Antibodies at Day 1
Description: Anti-PF-05231023 antibodies and neutralizing antibodies were analyzed only for participants who received PF-05231023 as per planned analysis. One sample at Day 1 was inadvertently tested for neutralizing antibody even though the corresponding anti-PF-05231023 antibody was negative.
Time Frame: Day 1
Population: Safety Analysis Set included all participants who receive at least 1 dose of study medication. Here "n" signifies those participants who were evaluable for this measure at specified time-points for each arm, respectively
Measure: Number; unit: participants
Arm/Group | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 21 | 21 | 22 | 21
participants
  Anti-PF- 05231023 Antibodies (n=21, 21, 22, 21) | 0 | 0 | 0 | 0
  Neutralizing Antibodies (n=0, 0, 0, 1) | NA — Data was not analyzed as none of the participant in this arm was evaluable for neutralizing antibody. | NA — Data was not analyzed as none of the participant in this arm was evaluable for neutralizing antibody. | NA — Data was not analyzed as none of the participant in this arm was evaluable for neutralizing antibody. | 0

36. Primary Outcome: Number of Participants With Anti-PF-05231023 Antibodies and Neutralizing Antibodies at Day 39
Description: Anti-PF-05231023 antibodies and neutralizing antibodies were analyzed only for participants who received PF-05231023 as per planned analysis. One sample at Day 39 was inadvertently tested for neutralizing antibody even though the corresponding anti-PF-05231023 antibody was negative.
Time Frame: Day 39
Population: Safety analysis set included all participants who received at least 1 dose of study medication. Here "n" signifies those participants who were evaluable for specified antibodies for each arm, respectively and "N" (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 19 | 18 | 14 | 19
participants
  Anti-PF- 05231023 Antibodies (n=19, 18, 14, 19) | 0 | 0 | 0 | 1
  Neutralizing Antibodies (n=0, 0, 1, 1) | NA — Data was not analyzed as none of the participant in this arm was evaluable for neutralizing antibody. | NA — Data was not analyzed as none of the participant in this arm was evaluable for neutralizing antibody. | 0 | 0

37. Primary Outcome: Number of Participants With Anti-PF-05231023 Antibodies and Neutralizing Antibodies at Day 49
Time Frame: Day 49
Population: as for outcome 36
Measure: Number; unit: participants
Arm/Group | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 19 | 18 | 14 | 19
participants
  Anti-PF- 05231023 Antibodies (n=19, 18, 14, 19) | 0 | 1 | 0 | 1
  Neutralizing Antibodies (n=0, 2, 0, 1) | NA — Data was not analyzed as none of the participant in this arm was evaluable for neutralizing antibody. | 1 | NA — Data was not analyzed as none of the participant in this arm was evaluable for neutralizing antibody. | 0

38. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of PF-05231023 After Single Dose
Description: AUCtau was calculated for the intact C-terminus and N-terminus PF-05231023 from the concentration-time data using standard non-compartmental method. Only participants who received PF-05231023 were to be analyzed for this outcome measure.
Time Frame: 0 (pre-dose), 0.5 (end of infusion), 1, 2.5, 3.5, 5.5, 9.5, 11.5 hours after start of infusion on Day 1, Day 4, 0 hours (pre-dose) on Day 8
Population: Pharmacokinetic (PK) parameter analysis set included all participants randomized and treated who had at least 1 of the PK parameters of interest. Here "N" (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Geometric Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 20 | 21 | 17 | 20
nanogram*hour per milliliter (ng*hr/mL)
  PF-05231023 C-Terminus | 108100 (41048) | 206200 (107110) | 376600 (134870) | 475600 (99316)
  PF-05231023 N-Terminus | 376100 (111420) | 693400 (214250) | 1508000 (253030) | 2004000 (405880)

39. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-05231023 After Single Dose
Description: Tmax was calculated for the intact C-terminus and N-terminus PF-05231023 from the concentration-time data using standard non-compartmental method. Only participants who received PF-05231023 were to be analyzed for this outcome measure.
Time Frame: 0 (pre-dose), 0.5 (end of infusion), 1, 2.5, 3.5, 5.5, 9.5, 11.5 hours after start of infusion on Day 1, Day 4, 0 hour (pre-dose) on Day 8
Population: PK parameter analysis set included all participants randomized and treated who had at least 1 of the PK parameters of interest.
Measure: Median (Full Range); unit: hours
Arm/Group | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 21 | 21 | 21 | 21
hours
  PF-05231023 C-Terminus | 0.5 [0.5 to 1.0] | 0.5 [0.5 to 11.5] | 0.5 [0.5 to 3.4] | 0.5 [0.5 to 1.03]
  PF-05231023 N-Terminus | 1.0 [0.5 to 5.6] | 1.0 [0.5 to 11.5] | 1.0 [0.5 to 9.5] | 1.0 [0.5 to 3.5]

40. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-05231023 After Single Dose
Description: Cmax was calculated for the intact C-terminus and N-terminus PF-05231023 from the concentration-time data using standard non-compartmental method. Only participants who received PF-05231023 were to be analyzed for this outcome measure.
Time Frame: as for outcome 39
Population: as for outcome 39
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 21 | 21 | 21 | 21
nanogram per milliliter (ng/mL)
  PF-05231023 C-Terminus | 7983 (2000) | 15250 (3672) | 32980 (7944) | 48320 (8376)
  PF-05231023 N-Terminus | 8881 (1743) | 16800 (4740) | 31750 (5134) | 44470 (8516)

41. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of PF-05231023 After Last Dose
Description: as for outcome 38
Time Frame: 0 (pre-dose), 0.5 (end of infusion), 1, 2.5, 3.5, 4.5 hours after start of infusion on Day 22, Day 24, 25, 29
Population: PK parameter analysis set included all participants randomized and treated who had at least 1 of the PK parameters of interest. Here "N" (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 19 | 18 | 15 | 19
ng*hr/mL
  PF-05231023 C-Terminus | 76520 (26169) | 136200 (34051) | 301200 (71897) | 424700 (97424)
  PF-05231023 N-Terminus | 467700 (136600) | 855500 (269920) | 1860000 (434690) | 2326000 (433010)

42. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-05231023 After Last Dose
Description: as for outcome 39
Time Frame: 0 (pre-dose), 0.5 (end of infusion), 1, 2.5, 3.5, 4.5 hours after start of infusion on Day 22, Day 24, 25, 29, 39, 49
Population: as for outcome 41
Measure: Median (Full Range); unit: hours
Arm/Group | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 20 | 18 | 16 | 19
hours
  PF-05231023 C-Terminus | 0.55 [0.50 to 1.02] | 0.53 [0.45 to 1.00] | 0.79 [0.48 to 3.50] | 1.00 [0.50 to 1.00]
  PF-05231023 N-Terminus | 1.00 [0.50 to 4.55] | 1.00 [0.48 to 4.50] | 1.00 [0.50 to 4.50] | 1.00 [0.50 to 4.52]

43. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-05231023 After Last Dose
Description: as for outcome 40
Time Frame: 0 (pre-dose), 0.5 (end of infusion), 1, 2.5, 3.5, 4.5 hours after start of infusion on Day 22, Day 24, 25, 29, 39, 49
Population: as for outcome 41
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 20 | 18 | 16 | 19
ng/mL
  PF-05231023 C-Terminus | 7697 (1622) | 14450 (3428) | 29610 (5300) | 42260 (7419)
  PF-05231023 N-Terminus | 9981 (3406) | 16900 (3279) | 33140 (9119) | 48090 (17688)

44. Secondary Outcome: Accumulation Ratio for Area Under the Curve From Time Zero to End of Dosing Interval (Rac) of PF-05231023
Description: Rac was obtained from AUCtau after last dose (Day 22) divided by AUCtau after single dose (Day 1). Rac was calculated for the intact C-terminus and N-terminus PF-05231023 from the concentration-time data using standard non-compartmental method. Only participants who received PF-05231023 were to be analyzed for this outcome measure.
Time Frame: 0 (pre-dose), 0.5 (end of infusion ), 1, 2.5, 3.5, 5.5, 9.5, 11.5 hours after start of infusion on Day 1; Day 4, 0 hour (pre-dose) on Day 8; 0 (pre-dose), 0.5 (end of infusion), 1, 2.5, 3.5, 4.5 hours after start of infusion on Day 22; Day 24, 25, 29
Population: as for outcome 41
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 19 | 18 | 15 | 19
ratio
  PF-05231023 C-Terminus | 0.70 (0.23) | 0.65 (0.20) | 0.79 (0.24) | 0.90 (0.17)
  PF-05231023 N-Terminus | 1.24 (0.20) | 1.28 (0.31) | 1.25 (0.15) | 1.16 (0.15)

45. Secondary Outcome: Accumulation Ratio for Maximum Observed Plasma Concentration (Rac,Cmax) of PF-05231023
Description: as for outcome 44
Time Frame: 0 (pre-dose),0.5(end of infusion), 1, 2.5, 3.5, 5.5, 9.5, 11.5 hours after start of infusion on Day 1; Day 4, 0 hour (pre-dose) on Day 8; 0 (pre-dose), 0.5 (end of infusion), 1, 2.5, 3.5, 4.5 hours after start of infusion on Day 22; Day 24,25,29,39,49
Population: as for outcome 41
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 20 | 18 | 16 | 19
ratio
  PF-05231023 C-Terminus | 0.93 (0.12) | 0.96 (0.20) | 0.89 (0.23) | 0.89 (0.22)
  PF-05231023 N-Terminus | 1.13 (0.27) | 1.04 (0.17) | 1.04 (0.33) | 1.10 (0.74)

46. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin) of PF-05231023 After Last Dose
Description: Cmin was calculated for the intact C-terminus and N-terminus PF-05231023 from the concentration-time data using standard non-compartmental method. Only participants who received PF-05231023 were to be analyzed for this outcome measure.
Time Frame: 0 (pre-dose), 0.5 (end of infusion), 1, 2.5, 3.5, 4.5 hours after start of infusion on Day 22, Day 24, 25, 29, 39, 49
Population: as for outcome 41
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 20 | 18 | 16 | 19
ng/mL
  PF-05231023 C-Terminus | 0.0001000 (0.00000) | 0.0001000 (0.00000) | 0.0001000 (0.00000) | 0.0001866 (3.2348)
  PF-05231023 N-Terminus | 768.3 (405.33) | 1213 (585.54) | 3293 (1287.0) | 4182 (1646.7)

47. Secondary Outcome: Average Plasma Concentration (Cav ) of PF-05231023 After the Last Dose
Description: Cav was calculated for the intact C-terminus and N-terminus PF-05231023 from the concentration-time data using standard non-compartmental method. Only participants who received PF-05231023 were to be analyzed for this outcome measure.
Time Frame: 0 (pre-dose), 0.5 (end of infusion), 1, 2.5, 3.5, 4.5 hours after start of infusion on Day 22, Day 24, 25, 29, 39, 49
Population: as for outcome 41
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 19 | 18 | 15 | 19
ng/mL
  PF-05231023 C-Terminus | 455.8 (156.12) | 810.7 (203.85) | 1793 (426.65) | 2529 (581.04)
  PF-05231023 N-Terminus | 2783 (812.93) | 5091 (1605.8) | 11060 (2593.9) | 13840 (2574.9)

48. Secondary Outcome: Plasma Decay Half-Life (t1/2) of PF-05231023
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half. Half-Life was calculated for the intact C-terminus and N-terminus PF-05231023 from the concentration-time data using standard non-compartmental method. Only participants who received PF-05231023 were to be analyzed for this outcome measure.
Time Frame: 0 (pre-dose), 0.5 (end of infusion), 1, 2.5, 3.5, 4.5 hours after start of infusion on Day 22, Day 24, 25, 29, 39, 49
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 19 | 18 | 15 | 19
hours
  PF-05231023 C-Terminus | 7.6 (1.0) | 7.4 (1.3) | 7.4 (1.2) | 8.6 (3.5)
  PF-05231023 N-Terminus | 121.6 (16.5) | 119.3 (24.5) | 114.8 (12.5) | 114.6 (12.0)

49. Secondary Outcome: Apparent Clearance (CL) of PF-05231023
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body. CL was calculated for the intact C-terminus and N-terminus PF-05231023 from the concentration-time data using standard non-compartmental method. Only participants who received PF-05231023 were to be analyzed for this outcome measure.
Time Frame: 0 (pre-dose), 0.5 (end of infusion), 1, 2.5, 3.5, 4.5 hours after start of infusion on Day 22, Day 24, 25, 29, 39, 49
Population: as for outcome 41
Measure: Geometric Mean (Standard Deviation); unit: liter/hour (L/hr)
Arm/Group | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Number analyzed (Participants) | 19 | 18 | 15 | 19
liter/hour (L/hr)
  PF-05231023 C-Terminus | 0.33 (0.09) | 0.37 (0.08) | 0.33 (0.09) | 0.35 (0.08)
  PF-05231023 N-Terminus | 0.05 (0.02) | 0.06 (0.02) | 0.05 (0.01) | 0.06 (0.01)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | PF-05231023 25 mg | PF-05231023 50 mg | PF-05231023 100 mg | PF-05231023 150 mg
Serious Adverse Events (participants affected / at risk) | 1/22 | 2/21 | 0/21 | 1/22 | 0/21
Other Adverse Events (participants affected / at risk) | 11/22 | 15/21 | 10/21 | 12/22 | 12/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=22) | PF-05231023 25 mg (N=21) | PF-05231023 50 mg (N=21) | PF-05231023 100 mg (N=22) | PF-05231023 150 mg (N=21)
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=22) | PF-05231023 25 mg (N=21) | PF-05231023 50 mg (N=21) | PF-05231023 100 mg (N=22) | PF-05231023 150 mg (N=21)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 3 | 8
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 2
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Feeling cold (General disorders) | 0 | 1 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 1 | 0
Hunger (General disorders) | 0 | 1 | 0 | 0 | 2
Infusion site haematoma (General disorders) | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 1 | 0
Vessel puncture site haemorrhage (General disorders) | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood pressure diastolic increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0 | 0 | 0 | 0
Electrocardiogram ST segment abnormal (Investigations) | 0 | 1 | 0 | 0 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 1 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 1 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 1 | 1 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 1 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 1 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.